# INFORMED CONSENT TO TAKE PART IN CLINICAL RESEARCH STUDY AND AUTHORIZATION TO DISCLOSE HEALTH INFORMATION

**STUDY TITLE:** A Phase I Clinical Trial to Evaluate the Safety,

Tolerability, Pharmacokinetic Profiles and Efficacy of Oral BB102 Tablets in Patients with

Advanced Solid Tumors (the "Study")

**SPONSOR:** BroadenBio Co., Ltd. ("*Sponsor*")

PROTOCOL NO.: BB102-ST-I-02

**INVESTIGATOR:** 

SITE(S):

**STUDY PHONE NUMBER(S):** (24-hour number)

### TABLE OF CONTENTS

| TABLE OF CONTENTS | 2 |
|---|---|
| INTRODUCTION | |
| PURPOSE OF THE STUDY | 4 |
| HOW MANY PEOPLE WILL TAKE PART IN THE STUDY? | |
| WHO IS SPONSORING THIS STUDY? | |
| WILL OTHERS BE INVOLVED WITH THE CONDUCT OF THIS STUDY? | 5 |
| STUDY DRUG TO BE USED | |
| HOW LONG WILL THE STUDY LAST | |
| TO BE IN THE STUDY | |
| WHAT WILL HAPPEN DURING THE STUDY | |
| LIST OF STUDY PROCEDURES | |
| Screening (Day -28 to -1): | |
| Single-dose Period (for dose escalation trial only) | |
| Day 1 (D1) | |
| Day 2 (D2) | |
| Day 3 (D3) | |
| Day 4 (D4) | |
| Day 5 (D5) | |
| Multiple-dose Period (for dose escalation trial and dose expansion trial) | |
| Day 1 of Cycle 1 (C1D1): | |
| Day 8 of Cycle 1 (C1D8; time window for corresponding examination: ±1 day): | |
| Day 15 of Cycle 1 (C1D15; time window for corresponding examination: ±1 day): | |
| Day 21 of Cycle 1 (C1D21; time window for corresponding examination: ±1 day): | |
| End of study treatment visit (EOT; within 7 days after the last dose) | |
| Safety Follow-up Visits (28 days (±7 days) after the last dose) | |
| Subsequent Follow-up Visits [once every 8 weeks (#) days) after the last dose]: | |
| Unscheduled visit DRUG TREATMENTS DURING THE STUDY | |
| MAY I CONTINUE TO TAKE MEDICATIONS THAT I TAKE? | |
| POSSIBLE SIDE EFFECTS AND RISKS OF THE STUDY DRUG | |
| RISKS OF THE STUDY DRUG | |
| Other Risks | |
| Reproductive Risks | |
| Future Risks | |
| POSSIBLE BENEFITS OF THE STUDY | 2.2 |
| WHAT OTHER CHOICES DO I HAVE | |
| CONFIDENTIALITY | |
| LEGAL RIGHTS | |
| PARTICIPATION IN THE STUDY | |
| CAN I LEAVE THE STUDY EARLY? | |
| NEW FINDINGS | |
| WILL IT COST ANYTHING TO BE IN THIS STUDY ? | |
| IS THE STUDY DOCTOR PAID FOR CONDUCTING THIS STUDY? | |
| WHAT IF I GET HURT OR SICK WHILE I AM IN THE STUDY? | |

| PAYMENT FOR BEING IN THE STUDY | 26 |
|---|---|
| THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED | |
| CONSENT | 27 |
| What is a consent form? | 27 |
| What is an Institutional Review Board (IRB)? | |
| Advarra IRB, the IRB for this Study | |
| AGREEMENT TO BE IN THE STUDY | |
| PERSON OBTAINING CONSENT | 30 |
| AUTHORIZATION (PERMISSION) TO USE AND DISCLOSE YOUR HEALTH | |
| INFORMATION FOR RESEARCH PURPOSES | 31 |
| A.Purpose of this form | 31 |
| B.What health information will be obtained, used or disclosed? | |
| C.Who may use and disclose your health information? | 31 |
| D.Who may receive or use the information? | 32 |
| E. What is the purpose of this research Study and how will my health information be | |
| utilized in the Study ? | 32 |
| F.Do I have to sign and date this authorization form? | 33 |
| G.If I sign and date, can I cancel my permission or withdraw from the research Study | later? |
| | 33 |
| H.When will my Authorization expire? | 33 |
| I. Will access to my medical record be limited during the research Study? | 33 |

### INTRODUCTION

The purpose of this informed consent form ("*ICF*" or "consent form") is to help you decide if you want to take part in this Study.

You are being asked to volunteer for a research Study. Please read this consent form carefully and ask questions as many as you need to decide if you would like to participate in this Study. This form may contain words or information that you do not understand. Please ask the Study doctor and Study Staff to explain anything you do not understand. You should also consider talking with family members or your primary care doctor.

Before you may take part in the Study, you will be asked to sign and date this consent form. You will be given a signed and dated copy to take with you. If you do not sign this consent form, you cannot participate in the Study. Signing this form does not mean that you can take part in the Study. If your Study doctor believes you are a good candidate, you will have a screening visit to see if you are eligible to be in this Study.

It is important to remember that your participation in the Study is voluntary. Even after you have signed this consent form, you can change your mind at any time and for any reason and stop being in the Study. There will be no penalty or loss of benefits to which you are otherwise entitled if you choose not to participate in this Study or withdraw from the Study.

If you do choose to stop being in the Study, you must notify the site staff and you do not need to state the reason for your withdrawal. As noted above, your withdrawal can take place at any time, but it will not impact medical information and samples/specimens that have been used up until the effective date of your withdrawal.

The Study doctor is being paid by the Sponsor, BroadenBio Co., Ltd., to conduct this Study.

You must be honest and complete in providing your medical history. Giving false, incomplete, or misleading information about your medical history, including past and present drug use, could lead to your removal from this research study, and may cause you very serious health problems.

### PURPOSE OF THE STUDY

This Study is an investigational clinical Study. This Study involves receiving an experimental drug referred to as BB102. In this consent form, BB102 is also called the Study Drug. 'Experimental' or "Investigational" means that the Study Drug is currently being tested and has not been approved by the United States (U.S.) Food and Drug Administration (FDA) or any other health care regulatory authority in other countries.

BB102 is a novel small molecular drug being developed as a potential therapy for the treatment of advanced solid tumors. This study consists of a dose escalation trial and an expansion trial, both of which are designed as multi-center and open-label trials.

This study is being conducted to evaluate the safety (side effects and laboratory values) and tolerability (how well you tolerate the side effects) of Study Drug, and to determine the MTD (maximum tolerated dose), or recommended phase II dose (RP2D). Meanwhile, the study will explore the preliminary anti-tumor activity of Study Drug in expansion phase (dose expansion phase). This Study will also assess the "PK" (which means the amount of Study drug that is in your blood and how fast your body absorbs, metabolizes and eliminates the Study drug from your body).

### HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

The Study will include 2 parts.

Dose escalation phase: Approximately 19-42 subjects are expected to be enrolled. The participants will be divided into 6 dosing groups.

Dose expansion phase: Up to 12-36 subjects will be enrolled in each expansion arm, based on the safety, tolerability, PK and efficacy data obtained in previous trials, 1 to 3 appropriate doses (e.g., 100 mg QD, 160 mg QD, and 240 mg QD) will be selected for the expansion trial.

### WHO IS SPONSORING THIS STUDY?

BroadenBio Co., Ltd., the sponsor of this Study, is the company that designed the Study and is the company that makes the Study Drug. BroadenBio Co., Ltd., is also called the *Sponsor* in this consent form

### WILL OTHERS BE INVOLVED WITH THE CONDUCT OF THIS STUDY?

Yes, the Sponsor has or will hire others to assist with conducting and managing the Study including Study sites such as the site that made you aware of this investigational clinical Study opportunity and other vendors in connection with this Study.

### STUDY DRUG TO BE USED

The Study Drug, BB102, is given as an oral administration (take the medicine by your mouth) tablet.

### HOW LONG WILL THE STUDY LAST

Dose escalation phase including: Screening Period, within 28 days; Single-dose Period, 5 days; Multiple-dose Period, 21 days/cycle; End of treatment visit (EOT) Period, within 7 days after the last dose; Safety follow-up visit Period, on Day  $28 \pm 7$  days after final dose of Study drug; Subsequent Follow-up visit Period, every 8 weeks  $\pm 7$  days.

Dose expansion phase including: Screening Period, within 28 days; Multiple-dose Period, 21 days/cycle; End of treatment visit (EOT) Period, within 7 days after the last dose; Safety follow-up visit Period, on Day  $28 \pm 7$  days after final dose of Study drug; Subsequent Follow-up visit Period, every 8 weeks  $\pm 7$  days.

You are free to stop taking part in this Study at any time and you need to tell the doctor.

### TO BE IN THE STUDY

You must be male or female, aged  $\geq$  18 years old. You are being asked to take part in this investigational drug Study (dose escalation phase) only if the Study doctor has determined that you have histologically, cytologically confirmed or clinically confirmed advanced solid tumors, without available standard treatment, failed in standard treatment or cannot tolerate standard treatment. You are being asked to take part in this investigational drug Study (dose expansion phase) only if the Study doctor has determined that you have histologically or cytologically confirmed FGF19 or FGFR4 positive advanced primary HCC or other advanced solid tumors patients who without available standard treatment, failed in standard treatment or cannot tolerate standard treatment.

As a subject, you are responsible for following the Study directions, your Study doctor, and study staff. This includes returning promptly to your Study doctor's office for the overnight confinement period and reporting any changes in how you feel to the Study doctor or Study staff.

If you experience any illness or discomfort during the Study, you should notify your Study doctor or Study staff. Your Study doctor will then evaluate you to determine if you should continue the Study.

During this Study, you should notify any doctor who is taking care of you that you are taking part in a research Study that involves the use of this investigational treatment.

As a subject in this research Study, you are expected to:

- Ensure that you do not take part in any other research Study until you are done taking part in this research Study.
  - O Taking part in another Study before this one ends could affect the results of this Study. Your part in this research Study will immediately end if you decide to take part in another research Study.
- Contact the Study staff and ask questions as you think of them.
- Tell the Study doctor or Study staff, as soon as possible, if you change your mind about staying in the Study.

### WHAT WILL HAPPEN DURING THE STUDY

If you decide to take part in this Study and your Study doctor believes you are a suitable candidate, you will have a screening visit to determine if you are eligible to be in this Study. If you are eligible, you will be enrolled in the Study and begin receiving the Study Drug. Many tests associated with this Study are performed as part of your regular health care. You may be familiar with these tests. If not, please ask the Study staff to explain any tests you do not understand. You will have the following tests and procedures performed before, during and after you are treated with the Study Drug.

## LIST OF STUDY PROCEDURES Screening (Day -28 to -1):

Before the Study starts, if you decide that you would like to participate in this Study, you will be asked to sign this consent form. Then you will need to have the following examinations, tests, and procedures within 28 days before the treatment to determine if you can take part in the Study (this is called the screening evaluation).

- Collection of your demographic information (age, gender, race and ethnicity)
- Collection of your medical history and medication history
- Hematology test will be performed. It should be completed within 7 days prior to the first dose, and abnormal test parameters with clinical significance can be re-tested once within 7 days as needed.
- Urinalysis will be performed. It should be completed within 7 days prior to the first dose, and abnormal test parameters with clinical significance can be re-tested once within 7 days as needed.
- Stool routine will be performed. It should be completed within 7 days prior to the first dose, and abnormal test parameters with clinical significance can be re-tested once within 7 days as needed.
- Blood biochemistry test will be performed (including Liver function, Renal function, Blood lipids, Electrolytes, Cardiac function and Blood glucose). It should be completed within 7 days prior to the first dose, and abnormal test parameters with clinical significance can be re-tested once within 7 days as needed.
- Coagulation test will be performed. It should be completed within 7 days prior to the first dose, and abnormal test parameters with clinical significance can be re-tested once within 7 days as needed.
- Vital signs test will be performed, including body temperature, blood pressure, heart rate, and respiration. It shoul be completed following the visit time window.
- 12-lead ECG measurements will be performed after resting in supine position. It shoul be completed following the visit time window.
- Physical examination will be performed by organ and system, including body height, body weight, body mass index (BMI), general condition, nervous system, head and neck, lymph nodes, skin, mucosa, chest, abdomen, four limbs and spine.
- ECOG assessment will be performed.
- Pregnancy-related test will be performed.
- Echocardiography (LVEF) test will be performed.
- Serum etiology tests will be performed, including HIV-Ab, hepatitis B surface antigen (HBsAg), HBV-DNA (as needed), hepatitis C virus antibody (HCV-Ab) and HCV-RNA (as needed). It should be completed within 14 days prior to the first dose.
- Tumor assessment will be performed. If you received a CT/MRI or other radiological examinations within 4 weeks prior to the first dose and has not received any anti-tumor therapy since this tumor assessment, and at the investigator's discretion, the tumor assessment can be performed according to RECIST v1.1, this examination result can be used as baseline tumor assessment result (repeated examination is not necessary).
- Biomarker detection will be performed.

- AE will be recorded.
- Inpatient nutrition assessment (NRS-2002) will be assessed as needed.
- The inclusion/exclusion criteria will be reviewed.

## Single-dose Period (for dose escalation trial only) Day 1 (D1)

The following procedures will be performed:

- Vital signs test will be performed, including body temperature, blood pressure, heart rate and respiration. For D1, it will be measured within 1 h pre-dose and at 10 h (± h) post-dose on D1. If there are corresponding clinical symptoms at other time, vital signs should also be measured, and the data should be recorded.
- 12-lead ECG measurements will be performed after resting in supine position, and the data (PR, QRS, QT and QTcF) will be recorded. For D1, it will be measured within 1 h predose and at 10 h (±1 h) post -dose on D1. If there are corresponding clinical symptoms at other time, ECG should also be performed, the data should be recorded, and the ECG results should be kept.
- Study drug administration will be performed.
- PK blood will be collected (within 0.5 h (0 h) before single-dosing and 1 h (\pm \text{min}), 2 h (\pm \text{min}), 4 h (\pm \text{0 min}), 6 h (\pm \text{0 min}), 8 h (\pm \text{0 min}), 10 h (\pm \text{0 min}) after dosing).
- Blood will be collected for metabolite identification.
- AE will be recorded.
- DLT evaluation will be performed.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### Day 2 (D2)

The following procedures will be performed:

- PK blood will be collected (24 h±1 h after dosing).
- Blood will be collected for metabolite identification.
- AE will be recorded.
- DLT evaluation will be performed.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### **Day 3 (D3)**

- Vital signs test will be performed, including body temperature, blood pressure, heart rate, and respiration. Follow the visit time window. If there are corresponding clinical symptoms at other time, vital signs should also be measured, and the data should be recorded.
- 12-lead ECG measurements will be performed after resting in supine position, following the visit time window. If there are corresponding clinical symptoms at other time, ECG should also be performed, the data should be recorded.
- PK blood will be collected (48 h±1 h after dosing).
- Blood will be collected for metabolite identification.
- AE will be recorded.
- DLT evaluation will be performed.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### Day 4 (D4)

The following procedures will be performed:

- PK blood will be collected (72 h±2 h after dosing).
- Blood will be collected for metabolite identification.
- AE will be recorded.
- DLT evaluation will be performed.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### Day 5 (D5)

- Hematology test will be performed.
- Urinalysis will be performed.
- Stool routine will be performed.
- Blood biochemistry test will be performed.
- Coagulation test will be performed.
- Vital signs test will be performed, including body temperature, blood pressure, heart rate, and respiration. Follow the visit time window. If there are corresponding clinical symptoms at other time, vital signs should also be measured, and the data should be recorded.
- 12-lead ECG measurements will be performed after resting in supine position, following the visit time window. If there are corresponding clinical symptoms at other time, ECG should also be performed, the data should be recorded.
- Physical examination will be performed per organ and system, and a simple physical
  examination will be performed at this visit, including but not limited to weight, BMI,
  general condition, skin, and any abnormal signs of concern at the investigator's
  discretion.

- ECOG assessment will be performed.
- PK blood will be collected (96 h±2 h after dosing).
- Blood will be collected for metabolite identification.
- AE will be recorded.
- DLT evaluation will be performed.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

## Multiple-dose Period (for dose escalation trial and dose expansion trial) Day 1 of Cycle 1 (C1D1):

The following procedures will be performed:

- Vital signs will be assessed, including body temperature, blood pressure, heart rate and respiration. For C1D1, it will be measured within 1 h pre-dose and at 10 h (± h) post dose on C1D1. If there are corresponding clinical symptoms at other time, vital signs should also be measured, and the data should be recorded.
- 12-lead ECG measurements will be performed. For C1D1, it will be measured within 1 h pre-dose and at 10 h (± h) post -dose on C1D1. If there are corresponding clinical symptoms at other time, ECG should also be performed, the data should be recorded, and the ECG results should be kept.
- Study drug administration will be performed.
- Dispensing diary cards and drugs will be performed.
- PK blood will be collected (within 0.5 h pre-dose).
- AE will be recorded.
- DLT evaluation will be performed.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### Day 8 of Cycle 1 (C1D8; time window for corresponding examination: $\pm 1$ day):

The following procedures will be performed:

You will be contacted via phone for survival status every 6 weeks  $\pm 7$  days post disease progression or starting new anti-tumor therapies until death, withdrawal of informed consent, lost to follow up, study termination by the sponsor or 12 months after the last dose of the study drug, whichever comes first

- Hematology test will be performed, and existing laboratory test results within 48 hours are acceptable.
- Urinalysis will be performed, and existing laboratory test results within 48 hours are acceptable.
- Stool routine test will be performed, and existing laboratory test results within 48 hours are acceptable.
- Blood biochemistry test will be performed (including Liver function, Renal function, Blood lipids, Electrolytes, Cardiac function and Blood glucose), and existing laboratory test results within 48 hours are acceptable.

- Coagulation test will be performed, and the existing laboratory test results within 48 hours are acceptable.
- Vital signs will be assessed, including body temperature, blood pressure, heart rate, and respiration, following the visit time window. If there are corresponding clinical symptoms at other time, vital signs should also be measured, and the data should be recorded.
- 12-lead ECG measurements will be performed after resting in supine position, following the visit time window. If there are corresponding clinical symptoms at other time, ECG should also be performed, the data should be recorded, and the ECG results should be kept.
- Physical examination will be performed per organ and system, including but not limited to weight, BMI, general condition, skin, and any abnormal signs of concern at the investigator's discretion.
- Study drug administration will be performed.
- PK blood will be collected (within 0.5 h pre-dose).
- AE will be recorded.
- DLT evaluation will be performed.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### Day 15 of Cycle 1 (C1D15; time window for corresponding examination: ±1 day):

- Hematology test will be performed, and existing laboratory test results within 48 hours are acceptable.
- Urinalysis will be performed, and existing laboratory test results within 48 hours are acceptable.
- Stool routine test will be performed, and existing laboratory test results within 48 hours are acceptable.
- Blood biochemistry test will be performed (including Liver function, Renal function, Blood lipids, Electrolytes, Cardiac function and Blood glucose), and existing laboratory test results within 48 hours are acceptable.
- Coagulation test will be performed, and the existing laboratory test results within 48 hours are acceptable.
- Vital signs will be assessed, including body temperature, blood pressure, heart rate, and respiration, following the visit time window. If there are corresponding clinical symptoms at other time, vital signs should also be measured, and the data should be recorded.
- 12-lead ECG measurements will be performed after resting in supine position, following the visit time window. If there are corresponding clinical symptoms at other time, ECG should also be performed, the data should be recorded, and the ECG results should be kept.

- Physical examination will be performed per organ and system, including but not limited to weight, BMI, general condition, skin, and any abnormal signs of concern at the investigator's discretion.
- Study drug administration will be performed.
- Biomarker detection will be performed.
- PK blood will be collected (within 0.5 h pre-dose).
- AE will be recorded.
- DLT evaluation will be performed.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### Day 21 of Cycle 1 (C1D21; time window for corresponding examination: ±1 day):

- Hematology test will be performed, and existing laboratory test results within 48 hours are acceptable.
- Urinalysis will be performed, and existing laboratory test results within 48 hours are acceptable.
- Stool routine test will be performed, and existing laboratory test results within 48 hours are acceptable.
- Blood biochemistry test will be performed (including Liver function, Renal function, Blood lipids, Electrolytes, Cardiac function and Blood glucose), and existing laboratory test results within 48 hours are acceptable.
- Coagulation test will be performed, and the existing laboratory test results within 48 hours are acceptable.
- Vital signs will be assessed, including body temperature, blood pressure, heart rate, and respiration, following the visit time window. If there are corresponding clinical symptoms at other time, vital signs should also be measured, and the data should be recorded.
- 12-lead ECG measurements will be performed after resting in supine position, it will be performed within 0.5 h pre-dose and at 2 h (±5 min), 4 h (±5 min), 6 h (±20 min), 8 h (±30 min) and 24 h (±1 h, pre -dose on C2D1) post-dose. If there are corresponding clinical symptoms at other time, ECG should also be performed, the data should be recorded, and the ECG results should be kept.
- Physical examination will be performed per organ and system, including but not limited to weight, BMI, general condition, skin, and any abnormal signs of concern at the investigator's discretion.
- ECOG assessment will be performed.
- Pregnancy-related test will be performed. For women of childbearing potential, HCG will be tested.
- Echocardiography will be performed (LVEF). During treatment, echocardiography will be performed at the same frequency with tumor assessment, i.e., echocardiography will be performed at the end of the 1st cycle, and the time window is ± day after the end of the cycle.

- Study drug administration will be performed.
- Dispensing/collecting diary cards and drugs will be performed.
- Tumor assessment will be performed. A tumor assessment will be performed at the end of Cycle 1, for which the time window is the end of the cycle ± 1 day [if a subject's assessment result is complete response (CR), partial response (PR) or stable disease (SD), the subject can continue the treatment and continue to receive tumor assessments once every 2 cycles]. The radiological confirmation examination of CR or PR should be completed 4-8 weeks after the first evaluation of CR or PR.
- PK blood will be collected (within 0.5 h pre-dose and 1 h (⅓ min), 2 h (⅓ min), 4 h (⅓ 0 min), 6 h (⅓ 0 min), 8 h (⅓ 0 min), 10 h (⅓ 0 min) and 24 h (⅓ 0 min; collected before dosing on C2D1)).
- AE will be recorded.
- DLT evaluation will be performed.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### Day 1 of Cycle 2 (C2D1; time window for corresponding examination: $\pm 1$ day):

The following procedures will be performed:

- PK blood will be collected.
- AE will be recorded.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

## Starting from Cycle 2 treatment, on Day 21 of each cycle of treatment (CnD21; time window for corresponding examinations: \(\pma\) days):

- Hematology will be performed. Twice in Cycle 2, e.g., D14 and D21 of the cycle, with a time window of \(\precedut{\prece}\precedut{\precedut{\precedut{\precedut{\precedut{\prece}\precedut{\precedut{\precedut{\precedut{\prece}\precedut{\prece}\precedut{\precedut{\precedut{\precedut{\precedut{\prece}\pre
- Urinalysis will be performed. For Cycle 2-5, once at the end of each cycle, with a time window of \(\pm\) days; since Cycle 6, once at the end of every 2 cycles, with a time window of \(\pm\) days.
- Stool routine test will be performed. For Cycle 2-5, once at the end of each cycle, with a time window of \(\pm\) days; since Cycle 6, once at the end of every 2 cycles, with a time window of \(\pm\) days.
- Blood biochemistry will be performed. Twice in Cycle 2, e.g., D14 and D21 of the cycle, with a time window of \(\preceq\) days; for Cycles 3 to 5, once at the end of each cycle, with a time window of \(\preceq\) days; since Cycle 6, once at the end of every 2 cycles, with a time window of \(\preceq\) days.
- Coagulation will be performed. Twice in Cycle 2, e.g., D14 and D21 of the cycle, with a time window of \(\preceq\) days; for Cycles 3 to 5, once at the end of each cycle, with a time window of \(\preceq\) days; since Cycle 6, once at the end of every 2 cycles, with a time window of \(\preceq\) days.

- Vital signs assessment will be performed, including body temperature, blood pressure, heart rate, and respiration, in accordance with the visit time window (twice in Cycle 2, e.g., D14 and D21 of the cycle, with a time window of \(\pm\) days; for Cycles 3 to 5, once at the end of each cycle, with a time window of \(\pm\) days; since Cycle 6, once at the end of every 2 cycles, with a time window of \(\pm\) days). If there are corresponding clinical symptoms at other time, vital signs should also be measured, and the data should be recorded.
- 12-lead ECG measurements will be performed after resting in supine position, in accordance with the visit time window (twice in Cycle 2, e.g., D14 and D21 of the cycle, with a time window of Ⅎ days; for Cycles 3 to 5, once at the end of each cycle, with a time window of Ⅎ days; since Cycle 6, once at the end of every 2 cycles, with a time window of Ⅎ days). If there are corresponding clinical symptoms at other time, ECG should also be performed, the data should be recorded, and the ECG results should be kept.
- Physical examination will be performed per organ and system, and a simple physical examination will be performed at this visit, including but not limited to weight, BMI, general condition, skin, and any abnormal signs of concern at the investigator's discretion. Twice in Cycle 2, e.g., D14 and D21 of the cycle, with a time window of Ⅎ days; for Cycles 3 to 5, once at the end of each cycle, with a time window of Ⅎ days; since Cycle 6, once at the end of every 2 cycles, with a time window of Ⅎ days.
- ECOG assessment will be performed. For Cycle 2-5, once at the end of each cycle, with a time window of \(\precedut{\prece}\precedut{\precedut{\precedut{\precedut{\precedut{\prece}\precedut{\prec
- Pregnancy-related tests will be performed. For women of childbearing potential, HCG will be tested. Blood HCG pregnancy test at screening visit should be completed within 7 days prior to the first dose. For Cycle 2-5, once at the end of each cycle, with a time window of Ⅎ days; since Cycle 6, once at the end of every 2 cycles, with a time window of Ⅎ days.
- Echocardiography (LVEF) will be performed. During treatment, echocardiography will be performed at the same frequency with tumor assessment, i.e., after the end of the 1st cycle, echocardiography will be performed every 2 cycles with a time window of ≠ days from the end of every 2 cycles.
- Study drug administration will be performed.
- Dispensing/collecting diary cards and drugs will be performed.
- Tumor assessment will be performed. Tumor assessments will be performed once every 2 cycles after the end of Cycle 1, for which the time window is the end of every 2 cycles ± 7 days [if a subject's assessment result is CR, PR or SD, the subject can continue the treatment and continue to receive tumor assessments once every 2 cycles]. The radiological confirmation examination of CR or PR should be completed 4-8 weeks after the first evaluation of CR or PR.
- Biomarker detection will be performed.
- AE will be recorded.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### End of study treatment visit (EOT; within 7 days after the last dose)

The following procedures will be performed:

- Hematology test will be performed, and the existing laboratory test results within the visit time window are acceptable.
- Urinalysis will be performed, and the existing laboratory test results within the visit time window are acceptable.
- Stool routine test will be performed, and the existing laboratory test results within the visit time window are acceptable.
- Blood biochemistry test will be performed (including Liver function, Renal function, Blood lipids, Electrolytes, Cardiac function and Blood glucose), and the existing laboratory test results within the visit time window are acceptable.
- Coagulation test will be performed, and the existing laboratory test results within the visit time window are acceptable.
- Vital signs assessment will be performed, including body temperature, blood pressure, heart rate, and respiration, following the visit time window. If there are corresponding clinical symptoms at other time, vital signs should also be measured, and the data should be recorded.
- 12-lead ECG measurements will be performed after resting in supine position, following the visit time window. If there are corresponding clinical symptoms at other time, ECG should also be performed, the data should be recorded, and the ECG results should be kept.
- Physical examination will be performed per organ and system, and a simple physical examination will be performed at this visit, including but not limited to weight, BMI, general condition, skin, and any abnormal signs of concern at the investigator's discretion.
- ECOG assessment will be performed.
- Pregnancy-related tests will be performed. For women of childbearing potential, HCG will be tested. For men and women ≥60 years of age, a pregnancy-related test is not required.
- Echocardiography (LVEF) will be performed.
- Collecting diary cards and drugs will be performed.
- The investigator will determine whether a tumor assessment is required according to the condition. If a tumor assessment has been performed within 2 months prior to EOT, it is not necessary to repeat the tumor assessment at EOT visit. The radiological confirmation examination of CR or PR should be completed 4-8 weeks after the first evaluation of CR or PR.
- Biomarker detection will be performed.
- AE will be recorded.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### Safety Follow-up Visits (28 days (±7 days) after the last dose)

- Hematology test will be performed, and the existing laboratory test results within the visit time window are acceptable.
- Urinalysis will be performed, and the existing laboratory test results within the visit time window are acceptable.
- Stool routine test will be performed, and the existing laboratory test results within the visit time window are acceptable.
- Blood biochemistry test will be performed (including Liver function, Renal function, Blood lipids, Electrolytes, Cardiac function and Blood glucose), and the existing laboratory test results within the visit time window are acceptable.
- Coagulation will be performed, and the existing laboratory test results within the visit time window are acceptable.
- Anti-cancer therapy and survival information after study treatment discontinuation will be recorded
- AE will be recorded.
- Concomitant medications will be recorded.
- Inpatient nutrition assessment will be assessed as needed.

### Subsequent Follow-up Visits [once every 8 weeks (±7 days) after the last dose]:

The following procedures will be performed:

- Tumor assessment will be performed, during the subsequent follow-up visits once every 8 weeks (±7 days) after the last dose, a tumor assessment will be performed for the subjects who are assessed as having no tumor progression in the previous assessment. Tumor assessments will be performed on subjects whose tumor has not progressed in the last assessment until the subject is lost to follow-up, the subject dies, the subject starts new anti-tumor therapy, the subject requests to withdraw from the trial and refuses to continue follow-up, the research data collection had reached the cutoff date, the study site is early closed, the study is early terminated, or the study ends (whichever occurs first). The radiological confirmation examination of CR or PR should be completed 4-8 weeks after the first evaluation of CR or PR.
- Biomarker detection will be performed.
- Anti-cancer therapy and survival information after study treatment discontinuation: During the follow-up period following study treatment discontinuation, the anti-cancer therapy and survival information of all subjects will be recorded. During the follow-up period after the end of the study treatment, all subjects will be followed up for the survival period and the tumor treatment status will be recorded until the subject is lost to follow-up, the subject dies, the subject requests to withdraw from the trial and refuses to continue follow-up, the research data collection had reached the cutoff date, the study site is early closed, the study is early terminated, or the study ends (whichever occurs first).
- Inpatient nutrition assessment will be assessed as needed.

### **Unscheduled visit**

• Temporary visit may be conducted when clinically needed. Both the content and results of unscheduled visits should be recorded in the original medical record and eCRF.

• In addition to the safety test items specified in the protocol, additional safety test items may be measured as necessary.

• Inpatient nutrition assessment will be assessed as needed.

### DRUG TREATMENTS DURING THE STUDY

The Study Drug will be given to you as tablets. In the Study, you will be asked to take a specific number of tablets by mouth daily in fasting state at the same medication time. You should take the Study Drug as instructed by the Study doctor and Study staff. You will be asked to return all used and unused bags of your Study Drug.

### MAY I CONTINUE TO TAKE MEDICATIONS THAT I TAKE?

Some medicines and over the counter drugs, including herbal supplements, may affect the way your body uses or gets rid of the Study Drug. Therefore, it is very important that you let the Study staff know about all the medicines and any over the counter drugs, including herbal supplements that you may be taking. Do not start taking something new during the Study without discussing it with the Study staff first.

### POSSIBLE SIDE EFFECTS AND RISKS OF THE STUDY DRUG

You must tell the Study doctor or Study staff about all side effects that you have. You must be honest about your side effects or it may not be safe for you to stay in the Study. Because the Study Drug is investigational drug, all of its side effects may not be known. There may be rare and unknown side effects. Some of the side effects may be life-threatening.

There are risks, discomforts, and inconveniences when taking part in any research Study. You should talk with the Study doctor if you have any questions.

Please tell the Study doctor or Study staff right away if you have any problems with your health or the way you feel after you sign and date this consent, whether or not you think these problems are related to the Study treatment. If you are not honest about your side effects, it may not be safe for you to stay in the Study.

### RISKS OF THE STUDY DRUG

The known or anticipated risks and discomforts associated with participating in the Study are described below. Throughout the Study, the experience and safety of the Study subjects will be closely monitored. You will be informed if changes are made to the Study and you may be asked to sign an updated version of this consent form.

### **Side Effects of the Drugs in this Study**

This is the first Study where the Study Drug is being given to humans. You may have side effects while participating in this Study. Like all medicines that are taken, everyone may have different side effects from the Study Drug.

 Side effects may be serious and/or life-threatening and may result in death. You should immediately tell your Study doctor or Study staff if you think you are having any side effects.

• Side effects can be long lasting or may never go away. If side effects from the Study Drug last for a long time, these long-lasting side effects could prevent you from getting different treatments in the future.

The study drug, BB102 has not been given to humans before; therefore, the potential side effects that could occur with BB102 in this Study cannot be predicted. All of the expectations concerning possible safety risks are based on laboratory and animal studies. The nonclinical toxicology studies have shown that BB102 was well tolerated in both SD rats and Beagle dogs. Based on the integrated toxicological findings in SD rats and Beagle dogs, the main toxic reactions which were related to BB102 and needed to be focused on were listed as follows:

The 28-day repeat-dose toxicity study in SD rats showed no changes in ophthalmologic examinations, coagulation parameters, or urine parameters related to BB102 citrate. The increased TBIL and moderate periportal hepatocyte vacuolization in female animals in the ≥150 mg/kg/day dose groups were considered as adverse changes, and liver was considered as the main toxic target organ. The liver related adverse changes exhibited signs of recovery during the recovery phase.

The 28-day repeat-dose toxicity study in Beagle dogs showed no changes in ophthalmologic examinations, body temperature, blood pressure, coagulation parameters, or urine parameters related to BB102 citrate. The moderate diffuse hepatocyte vacuolation in the liver of female animals in  $\geq$ 100 mg/kg/day dose groups was considered as an adverse change, and liver was considered as the main toxic target organ. The liver related adverse changes had completely reversed during the recovery phase.

The safety data now available of similar small molecule inhibitors of FGFR4 (FGF401, BLU-554, and H3B-6527) show that anaemia, abdominal pain, nausea, vomiting, ascites, constipation, diarrhea, fatigue, oedema, pyrexia, ALT increased, AST increased, ALP increased, blood bilirubin increased, γ-glutamyltransferase increased, and decreased appetite, etc. are the main adverse events (AEs). Inhibition of the FGF19/FGFR4 signaling pathway by such products can lead to an increase in the expression of CYP7A1 (CYP7A1 is involved in the biosynthesis of bile acids), which thereby leads to an increase in bile acid synthesis beyond the metabolic capacity of the liver, leading to cholestasis and consequently triggering a series of adverse reactions.

### Other Risks

You will undergo tests and procedures as part of this Study, some of which may be associated with side effects or other risks. Side effects, risks or discomforts include:

- Uncommonly, complications from biopsies can be life threatening. As with any interventional procedure, other potentially serious complications from bleeding or organ damage may occur. These might require additional surgical intervention
- Blood Sampling
  - o You may experience pain or redness and/or bruising at the needle injection site. Although rare, localized clot formation and 4

infections may occur. Light-headedness and/or fainting may also occur during or shortly after the blood draw. If you feel faint, you should immediately lie down to avoid falling.

### Radiological exams (CT/PET scan, MRI)

- o CT scans: CT scans use X-ray radiation. Radiation has the potential to cause cancer or harm an unborn child. The amount of radiation you will receive during a CT scan is very low and most doctors agree that the benefits outweigh the risks. Some CT scans require you take a "contrast solution" either by mouth, through the rectum or by injection into a vein. Although rare, the contrast solution may cause an allergic reaction such as nausea, vomiting, itching, skin rash or in very rare instances a swelling of the throat and difficulty in breathing. If you feel any of these symptoms or an allergic reaction you must tell the Study staff immediately so that you can be treated quickly. You may experience discomfort from lying still in an enclosed space for a prolonged period.
- O PET/CT scan: Positron Emission Tomography/Computed Tomography Scanning is a procedure in which pictures are made of your body after a radioactive metabolic tracer has been given to you. The results of this scan will help determine the existence, location and extent of disease. This will help in choosing the most effective treatment. A small amount of radioactive metabolic tracer will be injected into your body via an intravenous catheter or needle placed in a vein in your arm. The Federal Drug Administration (FDA) has determined that this compound is safe and has approved this drug for certain procedures. PET/CT scans have been performed throughout the world using the same metabolic tracer and they have had no adverse side effects in subjects having this procedure. The dose or amount of radiation you will receive will be similar to that received during chest and abdomen x-ray examinations.
- Magnetic Resonance Imaging (MRI): MRI scans create images of the body using a magnet and radio waves. While the procedure is much like a CT scan, there is no radiation involved in an MRI exam. While no significant risks have been found from the use of MRI scans, you may be bothered by the MRI machine noise and by feelings of being closed in (claustrophobia).

The contrast agent you may receive is FDA-approved and used routinely for MRI exams. It contains a material called gadolinium.

 About 1 in 100 people may notice discomfort, tingling or warmth in the lips, metallic taste in the mouth, tingling in the arm, nausea, or headache. These symptoms go away quickly.

- There is a small risk of an allergic reaction to gadolinium. However, a severe allergic reaction occurs in less than one in 300,000 people.
- The placement of the needle (small plastic tube) to give you the gadolinium may cause minor pain, bruising and/or infection at the injection site.

People with severe kidney failure who receive gadolinium are at risk of developing Nephrogenic Systemic Fibrosis/Nephrogenic Fibrosing Dermopathy (NSF/NFD). This disease causes fibrosis (the formation of too much connective tissue in the skin and internal organs). This is a serious disease, which can result in death.

You should notify the Study team or MRI staff if:

- you are allergic to gadolinium
- you have kidney problems

### • Electrocardiogram (ECG)

o You may experience mild discomfort or redness at the site of lead (sticker) placement. This kind of reaction usually is temporary and goes away by itself when the patches are removed.

### • Allergic Reactions

o Rare or unknown side effects could possibly occur, including life-threatening reactions. As with any drug, it is possible that you could have an allergic reaction to the Study Drug, such as itching, skin rash, facial swelling, and an acute or sudden drop in blood pressure. The sudden drop in blood pressure may lead to shock with loss of consciousness and/or possible seizures, including the possibility of death. If any of the above symptoms of an allergic reaction occurs, seek medical attention immediately.

### Other Drugs

o Using too much of any drug (over the counter, prescription or illegal), herbs or supplements, at any time during the Study, without approval from your Study doctor, could result in serious or even life-threatening reactions. Specifically, you should not use any new medications or supplements without first checking with the Study doctor. These drugs affect the way your body uses the Study Drug. Therefore, it is very important that you let the Study staff know about all medicines and any over-the-counter medications including herbal supplements that you may be taking.

### **Reproductive Risks**

The risks of the Study Drug to pregnant women, unborn children, and breastfed babies are not known. No studies have been conudcted to specifically evaluate the impact of the Study Drug on fertility or reproductive functions in any genders. The effects of the Study Drug on fetus (unborn

baby) are unknown. If you are a man, and your partner becomes pregnant when you are being in this Study, potential unknown injury may occur to the fetus (unborn baby). Women cannot take part in this Study if they:

- Are pregnant or breastfeeding; or
- Think they might be pregnant or might become pregnant during the Study.

Before entering the Study, each person in this Study must agree with his or her Study doctor: (i) on the method(s) of birth control (described below) that he or she will use (and such methods may include a backup method of birth control) and (ii) how long he or she will use the birth control.

If you have been surgically sterilized or have been through menopause (discuss this with your Study doctor), you do not need to meet any contraception requirements to take part in this Study. Sterilization includes bilateral tubal ligation or bilateral oophorectomy or hysterectomy.

In order to participate in this Study, males of reproductive potential and females of childbearing potential must also agree to one of the following from the time of signing the ICF through the last dose of study drug:

- Total abstinence. Periodic abstinence methods (such as calendar method, ovulation method, symptom-body temperature method, post-ovulation method) are not allowed.
- One of the contraceptive methods with a failure rate of <1%:
  - Intrauterine device or intrauterine hormone release system with an annual failure rate of <1%;
  - Males undergo vasoligation;
  - Double barrier method: Condoms and/or occlusion caps (diaphragm or cervical cap/dome cap), spermicide (foam/gel/film/cream/suppository) barrier method should be used as supplementary measures

## Within 6 months after the last administration, you can also accept the following contraceptive methods:

- Reasonable combined use of oral/injection/transdermal hormonal contraceptives that can inhibit ovulation (including estrogen and progesterone);
- Reasonable use of progesterone-only oral/injection/transdermal hormonal contraceptives that can inhibit ovulation.

If you become pregnant, or you suspect that you are pregnant, while in this Study or within 6 months after the last dose, notify the Study doctor or Study staff at once. If you become pregnant while in the Study, the Study Drug will be stopped, and you will be immediately withdrawn from the Study. If the pregnancy has occurred within 6 months after the last dose, the Study doctor will follow the progress of your pregnancy, will refer you for obstetrical care if necessary, will request access to your and/or your infant's medical records and will report the outcome to the Sponsor.

The Sponsor has not set aside any funds to pay for any aspects of obstetric, child or related care and does not plan to pay for them.

For more information about risks and side effects, ask your Study doctor.

### **Future Risks**

Since the Study Drug may stay in your body for up to one month, it may interact with some new medicines that your doctor may give you. It is important for you to tell your doctor(s) that you were in this Study and took the Study Drug so that they may take this information into consideration for your future treatments.

### POSSIBLE BENEFITS OF THE STUDY

We hope that you will get personal medical benefit from taking part in this study, but we cannot be certain. These potential benefits could include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer. Because there is not much information about the drug's effect on your cancer, we do not know if you will benefit from taking part in this study, although the knowledge gained from this study may help others in the future who have cancer.

### WHAT OTHER CHOICES DO I HAVE

Currently available treatments for advanced solid tumors also include surgery and/or chemotherapy, or other existing anti-tumor drugs. In addition, you could take part in another study. You could discuss these other treatments with your doctor to decide whether you want to participate in this study.

### CONFIDENTIALITY

Certain people and organizations will need to see, copy, and use your health data so that they can do their part in the Study. They are called 'authorized users.' Authorized users will be given access to and may make copies of your health data. This health data may or may not include your name. It may be traced back to you even if it does not include your name.

To ensure that your information collected for this Study will be kept private, your name will not be used whenever possible. A code will be used instead of your name. All of your Study data will be kept in a secure location.

Authorized users may include:

- Representatives of BroadenBio Co., Ltd..
- Representatives of IRB (a Research Ethics Review Board that reviews this Study).
- The Food and Drug Administration (FDA) and other US governmental agencies.
- Government agencies to whom certain diseases (like HIV, hepatitis, and STDs) must be reported.
- Governmental agencies of other countries.
- Labs working with the Sponsor on this Study.
- Other authorized users

Your health data needs to be shared for the research and other reasons. Therefore, complete privacy of your health data cannot be promised. However, sharing your health data will be guided by professional standards and the law.

Information from this Study may be presented at meetings or published in medical journals. The information included at meetings or in journals will not include your name or information that can easily be traced back to you.

#### LEGAL RIGHTS

You will not lose any of your legal rights as a research subject by signing and dating this consent form.

### GETTING ANSWERS TO YOUR QUESTIONS OR CONCERNS ABOUT THE STUDY

You can ask questions about this consent form or the Study (before you decide to start the Study, at any time during the Study, or after completion of the Study). Questions may include:

- Who to contact in the case of a research-related injury or illness;
- Payment or compensation for being in the Study, if any;
- Your responsibilities as a Study subject;
- Eligibility to participate in the research;
- The Study doctor's or Study site's decision to exclude you from participation;
- Results of tests and/or procedures;
- Other questions, concerns, or complaints.

Contact the Study doctor or Study staff <u>listed on the first page of this form</u> with any questions, concerns or complaints.

## GETTING ANSWERS TO YOUR QUESTIONS ABOUT YOUR RIGHTS AS A RESEARCH SUBJECT

This Study has been reviewed by an Institutional Review Board (IRB). This Committee reviewed this Study to help ensure that your rights and welfare are protected and that this Study is carried out in an ethical manner.

For questions about your rights as a research subject, contact:

• By mail:

[IRB name and address]

- or call **toll free**: [Tel]
- or by **email**: [email]

Please reference the following number when contacting the Study Subject Adviser:

• call **toll free**: [Tel]

### PARTICIPATION IN THE STUDY

Your participation in this Study is voluntary. You may withdraw from the Study at any time. You do not have to be in the Study if you don't want to, and you can change your mind at any time. There will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled.

The Study doctor, the sponsor company, the FDA, or IRB may remove you from the Study at any time for the following reasons:

- If you do not follow the instructions of the Study doctor
- You become pregnant
- If it is discovered that you do not meet the Study requirements
- If the Study is cancelled
- If it becomes harmful to your health

If you leave the Study, or if you are taken out of the Study for any reason, you may be asked to return to the Study site for a final visit to have some end of Study evaluations or tests. If you leave the Study, no more information about you will be collected for this Study. However, all of the information you gave us before you left the Study will still be used.

### CAN I LEAVE THE STUDY EARLY?

If you agree to take part in the Study but then change your mind, you are free to withdraw your consent and stop taking part at any time without loss of benefits to which you are entitled.

If you decide to stop taking part in this Study, you must notify your Study doctor that you wish to stop. It will be necessary for you to return to the Study center for a final visit. During this Study visit, the Study staff will collect all Study -related supplies, and your Study doctor will assess your health before leaving the Study. You can also discuss with your Study doctor how to best continue your medical care. You may be asked to return to the Study center after the final visit for safety assessments and follow up.

If you choose to leave the Study early, you will not be able to withdraw any data that was collected about you prior to leaving the Study . This data will remain in the Study site.

### **NEW FINDINGS**

You will be told of any important new information that is learned during the course of this research Study that might affect your condition or your willingness to continue taking part in this Study. You may be asked to sign and date a new informed consent form.

### WILL IT COST ANYTHING TO BE IN THIS STUDY?

It is not expected of you to have any costs for taking part in this Study. Items related to the routine medical care that you would receive even if you did not take part in this Study will be

billed to you or your insurance company,that means your medical cares won't related to this Study but you may need to be billed.

If you have any cost-related questions or concerns, please ask your Study doctor or Study staff.

#### IS THE STUDY DOCTOR PAID FOR CONDUCTING THIS STUDY?

BroadenBio Co., Ltd., the sponsor of this Study, is providing financial support and material for this Study and is paying for the Study doctor to conduct this Study. Any questions you have about other financial arrangements between the sponsor and the Study doctor or other Study staff can be discussed with the Study doctor.

### WHAT IF I GET HURT OR SICK WHILE I AM IN THE STUDY?

If you become ill or are hurt while you are in the Study, get the medical care that you need right away. You should inform the healthcare professional treating you that you are participating in this Study.

If you suffer any side effect or injury, notify the Study doctor immediately so that you can receive appropriate medical treatment.

If you suffer any injury as a direct result of the Study procedures or the Study drug, and not due to the natural course of any underlying disease or the treatment process for such condition, and you have commercial or other non-governmental insurance benefits, reimbursement for all related costs of care will be sought first from your insurer or managed care plan.

If costs of care related to such an injury are not covered by your insurer or managed care plan, or are not covered by a Federal or State benefits program, the Sponsor will pay for reasonable and necessary medical expenses that are a direct result of the Study procedures or the Study drug, and not due to the natural course of any underlying disease or the treatment process for such condition. The Sponsor will not agree to pay for such expenses if you did not follow the directions of the Study doctor and/or the Study staff.

To pay these medical expenses, the Sponsor will need to know some information about you like your name, date of birth, and social security number or Medicare Health Insurance Claim Number. This is because the Sponsor has to check to see if you receive Medicare and if you do, report the payment it makes to Medicare. The Sponsor will not use this information for any other purpose. Neither the Sponsor nor the Study doctor will provide other compensation in the event of an injury. However, you are not precluded from seeking to collect compensation for injury related to malpractice, fault, or blame on the part of those involved in the research.

Please be aware that some insurance plans may not pay for research-related injuries. You should contact your insurance company for more information.

In no way does signing and dating this consent form waive your legal rights nor does it relieve the investigators, Sponsor or involved institutions from their legal and professional responsibilities.

### PAYMENT FOR BEING IN THE STUDY

| You will be paid if you are discharged on Day 1, or if you are discharged on Day, within days of the completion of your taking part in this research Study . No additional financial compensation will be provided. |
|---|
| If your taking part in this research Study is terminated for any other reason, you will receive compensation based on the visits and/or day* that you have completed (*you will not receive payment for partial days) as outlined above. |
| You may also be asked to participate as an alternate for this Study. To be considered an alternate you must meet all of the eligibility requirements. If you are an alternate, but do not receive Study medication, you will be compensated for each overnight stay and the time spent in the clinic the following morning. If you choose to leave before dosing is complete, you will not be considered as an alternate. If you do not meet the eligibility requirements, you will not be considered an alternate. |
| Please note: if you have a positive test for drug abuse (including alcohol and/or cotinine if applicable) after starting this Study, you will receive a maximum amount of \$ for your entire participation in this Study. No other compensation will be paid. |
| You will be issued a Clincard, which is a specially designed debit card for clinical research onto which your compensation funds will be loaded as appropriate. When your participation is completed, funds will be approved and loaded onto your card within three business days. Once the funds are loaded the funds will then be available for use at your discretion. You will be issued one card for the duration of your participation. You should bring your card to each Study visit. If your card is lost or stolen, you can contact customer service. There is a fee for replacement and it will take 7-10 days to receive by mail. If you prefer, a replacement card can |

Additionally, you will have the option to receive updates related to appointment reminders and payment reminders via text message and email message (Standard text messaging rates will apply). You will have the opportunity to opt-in to receive these messages, you are not required to provide your cell phone or email address to be enrolled in the Study or use a ClinCard. If you choose to receive messages and decide at a later date that you want to stop these messages, you will have the ability to opt-out.

Any demographic information collected is stored in a secure fashion and kept completely confidential.

be issued at the site for a fee of , which will be deducted from your balance.

In agreeing to participate in this Study, you will be acting as an independent contractor. Because payments made to you for participating in this Study will be reported to the IRS as income as required by law, you are required to provide your Social Security Number. No deductions for any state or federal withholding or any other similar taxes will be made. It is the responsibility of the subject to report this compensation on state and federal tax returns and for the payment of any taxes that are due on this compensation.

### THE REASON FOR INSTITUTIONAL REVIEW BOARDS AND INFORMED CONSENT

### What is a consent form?

The informed consent document contains information required by federal regulations. The informed consent document must be approved by an Institutional Review Board (IRB).

### What is an Institutional Review Board (IRB)?

An Institutional Review Board (IRB) is a group of people that reviews research studies. The main goal of this review is to protect the rights and well-being of the human subjects participating in research studies.

### Advarra IRB, the IRB for this Study

Advarra IRB is an IRB whose board members provide IRB services across the United States.

To meet the requirements of the law, the Advarra's IRB Boards currently include:

- Doctors
- Pharmacists
- Nurses
- Toxicologists (people who Study the harmful effects of chemicals)
- Other specialists
- Others who do not have a background in science/medicine

Do not sign and date this consent form unless you have had a chance to ask questions and have received answers to all of your questions. If you agree to participate in the Study, please sign and date this document and you will receive a signed and dated copy to take home with you. Your signature indicates:

- That you have read and understood the above information
- That you have discussed this Study with the person obtaining consent
- That you have had the opportunity to ask any questions you may have
- That all of your questions have been answered to your satisfaction
- That you have decided to take part voluntarily (of your free will) based on the information provided

• That a copy of this form has been given to you

Your signature also indicates that you authorize the release of your medical records related to this Study to the Sponsor, the Study center, Advarra IRB, the FDA, and other regulatory agencies for purposes related to the Study or the Study drug.

### AGREEMENT TO BE IN THE STUDY

This consent form contains important information to help you decide if you want to be in the Study . If you have any questions that are not answered in this consent form, ask one of the Study staff.

Please answer YES or NO to the following questions:

A. Is this document in a language you understand?

B. Do you understand the information in this consent form?

C. Have you been given enough time to ask questions and talk about the Study?

D. Have all of your questions been answered to your satisfaction?

E. Do you think you received enough information about the Study?

F. Do you volunteer to be in this Study of your own free will and without being pressured by the Study doctor or Study staff?

G. Do you agree to take part in this Study?

H. Do you understand that you can leave the Study at any time without giving a reason and without affecting your medical care?

I. Do you understand that your medical records from this Study may be reviewed by BroadenBio Co., Ltd. (Sponsor), and by government authorities?

| IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUESTIONS, |
|--------------------------------------------------------|
| OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QUESTIONS |
| YOU SHOULD NOT SIGN AND DATE THIS CONSENT FORM. |

| Printed Name of Adult Study Subject | | |
|-------------------------------------|-----------|------|
| | / | _ |
| Signature of Adult Study Subject | :<br>Date | Time |

### PERSON OBTAINING CONSENT

I attest that the requirements of the informed consent for the medical research project described in this form have been satisfied that I have discussed the research project with the subject and explained to him or her in nontechnical terms all of the information contained in this informed consent form, including any risks and side effects that may reasonably be expected to occur. I certify that the information provided was given in a language that was understandable to the subject. I further certify that I encouraged the subject to ask questions and that all questions asked were answered.

| Printed Name of Person Explaining Informed Consent | | |
|----------------------------------------------------|------|------|
| | / / | : |
| Signature of Person Explaining Informed Consent | Date | Time |

You will be given a signed and dated copy of this informed consent form to keep.

### AUTHORIZATION (PERMISSION) TO USE AND DISCLOSE YOUR HEALTH INFORMATION FOR RESEARCH PURPOSES

### A. Purpose of this form

State and federal privacy laws protect the privacy of your health information. Under the law, health information that includes identifiable participant information may not be used for research purposes unless you give written permission in advance. You do not have to sign and date this Authorization. If you do not sign and date this Authorization, you will not be allowed to take part in this research Study. Your decision not to sign and date this Authorization will not affect any other treatment, healthcare, enrollment in health plans or eligibility for benefits.

Your health information will only be used in accordance with this authorization form and the informed consent form and as required or allowed by law. Please read it carefully before signing and dating it.

### B. What health information will be obtained, used or disclosed?

Health information related to this Study may be used or disclosed in connection with this research Study. Health information shall mean information contained in your medical or other healthcare records. Health information may include, protected health information that can identify you. For example, it may include but not be limited to your name, mailing/email address, phone number, birthdate, medical record number and social security number. Health information collected in connection with this research Study may also be found in the following:

- Progress notes
- Personal questions
- Health and medication questions
- Vital signs measurement
- History and Physical exams
- Laboratory Reports
- Menstrual or menopausal status
- Pregnancy tests
- Electrocardiograms (ECGs)
- All research related information and Study data

### C. Who may use and disclose your health information?

The following parties are authorized to use and/or disclose your health information in connection with this research Study:

- The Principal Investigator
- BroadenBio Co., Ltd., and any other affiliates, subsidiaries, agents, contractors and related companies of BroadenBio Co., Ltd., as necessary
- Study doctor's Study staff

- SRC (Safety Review Committee)
- IRB

### D. Who may receive or use the information?

The parties listed in Section C above may disclose your health information to the following persons and organizations in connection with this research Study:

- Sponsor and/or its representatives, including affiliates, agents and contractors ("Sponsor");
- Contract Research Organization (CRO);
- Business associates working with the Sponsor on this research Study (for example, laboratories);
- Independent Review Boards (IRB) who oversee this research Study: Advarra IRB;
- The Office for Human Research Protections in the US Department of Health and Human Services;
- Federal and regulatory authorities (for example, United States Food and Drug Administration-FDA), including those outside of the United States.

## E. What is the purpose of this research Study and how will my health information be utilized in the Study?

Your information about you and your health, and information that may identify you is being collected for the purposes of the research Study . The Sponsor will use your information to check the safety and results of the research Study and to seek government approval of the Study drug in order to market the Study drug.

Regulatory authorities and the IRB may also review and copy your information to make sure that the research Study is done properly or for other purposes required by law.

The results of this research Study may also be presented at scientific or medical meetings or published in scientific journals. Your identity will not be disclosed in any of these meetings or publications.

Your information may also be used along with the medical information of others to make and keep a research database. The database will be used for follow-up or future research and/or statistical purposes regarding medical conditions such as yours.

Your information may also be transferred to other countries which may have different privacy laws

### F. Do I have to sign and date this authorization form?

You do not have to sign and date this authorization form. But if you do not, you will not be able to take part in this research Study and you will not be able to receive any research-related Study treatment.

Signing and dating the form is not a condition for receiving any medical care outside the Study.

## G. If I sign and date, can I cancel my permission or withdraw from the research Study later?

You are free to withdraw or cancel your permission regarding the use and disclosure of your health information (and to discontinue any other participation in the Study ) at any time. After any cancellation or withdrawal, your health information will no longer be used or disclosed in the research Study , except to the extent that the law allows us to continue using your information (for example, information necessary to maintain the integrity or reliability of the research). Any revocation will not be effective to the extent that we have already taken an action in reliance on your authorization. If you wish to cancel or withdraw your permission for the research use or disclosure of your health information in this research Study , you must provide written notice in advance.

If you cancel or withdraw (or stop participating) from the research Study and cancel and withdraw this Authorization, no new information will be collected for the research Study purposes unless the information concerns a side effect related to the research Study . If a side effect occurs, your entire medical record may be reviewed. All information that has already been collected for research Study purposes, and any new information about a side effect related to the Study , will be sent to the Study Sponsor.

Your information may be subject to re-disclosure by the recipients described above. If those recipients are not required by law to protect the privacy of the information, it would thus no longer be protected by this Authorization or by law.

### **H.** When will my Authorization expire?

This Authorization does not have an expiration date. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely.

### I. Will access to my medical record be limited during the research Study?

To maintain the scientific integrity of this research Study, you may not have access to any health information developed as part of this Study until the Study is completed. At that point, you would have access to such health information if it was used to make a medical or billing decision about you (for example, if it was included in your official medical record). If it is necessary for your care, your health information will be provided to you or your doctor.

### **AUTHORIZATION**

[Insert Company Name of CRO] is required by law to protect your health information. By signing and dating this document, you authorize [Insert Company Name of CRO] to use and/or disclose (release) your health information for this research Study. Those persons who receive your health information may not be required by federal privacy laws (such as the Privacy Rule) to protect it and may share your information with others without your permission, if permitted by laws governing them. You acknowledge that you have received a copy of this form.

| Printed Name of Adult Subject | |
|------------------------------------------------|------|
| Signature of Adult Subject | Date |
| Printed Name of Person Obtaining Authorization | |
| Signature of Person Obtaining Authorization | Date |